CLINICAL TRIAL: NCT00543166
Title: Sex Steroids in Sjögren's Syndrome: Effect of Substitution Treatment on Fatigue
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Helsinki (Other)
Collaborators: Göteborg University (Other); Uppsala University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: T101090002
Record Dates: First submitted 2007-10-09; First posted 2007-10-12 (Estimated); Last update posted 2007-11-05 (Estimated); Status verified 2007-10

CONDITIONS: Sjogren's Syndrome
Keywords: Sjögren's syndrome; fatigue; salivary gland; dehydroepiandrosterone
MeSH Terms: conditions — Sjogren's Syndrome; Fatigue | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2 (Placebo Comparator): 180 patients divided to two separate groups (each containing 90 patients). This study has a cross-over, wash-out design, which consists of two 4 month treatment period separated by a one month long wash-out period. During one treatment period the patient gets placebo and during one of the treatment periods the patient gets 50mg of dehydroepiandrosterone (DHEA) in the morning.
  Interventions: Drug: dehydroepiandrosterone

INTERVENTIONS:
Drug: dehydroepiandrosterone — 50 mg of dehydroepiandrosterone in the morning for 4 months in the treatment group.
  Other Names: DHEA

SUMMARY:
Our research contributes to the understanding of some of the basic biology of the salivary glands. The etiology and many of the pathomechanisms of Sjögren's syndrome are unknown. In particular, reasons for the female dominance, late age of onset, fatigue and the prominent involvement of exocrine glands are unknown. We hypothesize, due to the disease characteristics, that the primary target hit by the disease process is the secretory acinar cell and that this cell is particularly damaged in women due to insufficient support, normally provided by dehydroepiandrosterone and its intracrine processing.

DETAILED DESCRIPTION:
We hypothesize, due to the Sjögren's syndrome (SS) disease characteristics, that the primary target hit by the disease process is the secretory acinar cell and that this cell is particularly in women damaged due to insufficient support, normally provided by dehydroepiandrosterone and its intracrine processing. Dehydroepiandrosterone deficiency at the time of adrenopause seems to us as the more likely endocrine trigger than estrogen deficiency caused by menopause as androgens in general are considered to be protective against autoimmunity and estrogens to favor it. Acinar cell is normally responsible for the production of primary saliva. Acinar cell damage can lead to acinar cell apoptosis and loss. Normally this is compensated by division of the acinar cells in situ or, according to recent reports, perhaps rather by division and subsequent migration of one of the daughter cells into the acinar space and transdifferentiation of this intercalated ductal cell progenitor into mature acinar cell. In SS this remodeling seems to be impaired, perhaps for the same reason, which also leads to primary acinar cell damage. According to this hypothesis, the primary changes occur in the salivary glands and more specifically in the acinar cells, whereas immune activation and autoimmunity are secondarily activated against abnormally damaged acinar cells so that individuals with the "right" genetic background also produce SS-A and SS-B antibodies. The cause of the acinar cell damage may not be a direct, damaging stimulus, e.g. virus infection or irradiation damage, but rather lack of a supporting anabolic stimulus and inadequate maintenance of the acinar cell health leading to cytopathic acinar cell changes. In peri-menopausal women (who still produce some estrogens) this abnormal antigen release and processing from acinar cells, which reveals cryptic epitopes, together with autoimmunity enhancing effects of estrogens, may lead to the full picture of SS (Cutolo et al., 2004).

This neuroimmunoendocrine working hypothesis would explain many central disease characteristics, but does not provide a final answer to the mystery of this intriguing syndrome as the reasons for the insufficient production and generation of DHEA remain to be solved. We have done some preliminary studies to analyze this topic by mapping the signals of the extracellular matrix in the adrenal cortex, where the cells proliferate in the outer zone and subsequently migrate in a centripetal direction, during which phenotypic transition occurs from the outer zone (zona glomerulosa) cells producing aldosterone to the intermediate zone (zona fasciculata) cells producing glucocorticosteroids and finally to the inner zone (zona reticularis) cells producing DHEA. However, in this research project we have decided to totally focus on the salivary gland acinar cell-sex steroid interactions.

ELIGIBILITY:
Inclusion Criteria:

1. Primary SS according to the American-European consensus criteria
2. General Fatigue ≥14 calculated from MFI-20 (Multiple fatigue inventory-20 questionnaire; the value was based on a pilot study of 239 members of the Finnish SS patient association)
3. subnormal serum S-DHEAS values (the reference values were calculated based on a pilot study of 81 healthy women and 57 healthy men).

Exclusion Criteria:

1. Age <18 years or >80 years
2. prisoner
3. individuals not able to give their informed consent
4. history of breast cancer
5. history of uterus cancer
6. history of prostatic cancer
7. history of stroke or prothrombotic coagulation disorders
8. pregnant or lactating women
9. fertile patients without adequate prevention
10. difficult acne
11. a significant liver disease
12. patients with changes in their systemic medication taken for SS during the previous three months 13) patients taking more than 10 mg prednisolone per day

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2003-02; Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Fatigue | prospective

SECONDARY OUTCOMES:
Quality of life | prospective

CONTACTS AND LOCATIONS:
Overall Officials: Yrjö Konttinen, MD, PhD, Principal Investigator — Helsinki University Central Hospital, Helsinki, Finland
Locations (1):
- Department of Medicine, Helsinki University Central Hospital, Helsinki, Helsinki, Finland

REFERENCES:
- [Background] Laine M, Virtanen I, Salo T, Konttinen YT. Segment-specific but pathologic laminin isoform profiles in human labial salivary glands of patients with Sjogren's syndrome. Arthritis Rheum. 2004 Dec;50(12):3968-73. doi: 10.1002/art.20730. PMID 15593200
- [Background] Konttinen YT, Tensing EK, Laine M, Porola P, Tornwall J, Hukkanen M. Abnormal distribution of aquaporin-5 in salivary glands in the NOD mouse model for Sjogren's syndrome. J Rheumatol. 2005 Jun;32(6):1071-5. PMID 15940770
- [Background] Valtysdottir ST, Wide L, Hallgren R. Low serum dehydroepiandrosterone sulfate in women with primary Sjogren's syndrome as an isolated sign of impaired HPA axis function. J Rheumatol. 2001 Jun;28(6):1259-65. PMID 11409117
- [Result] Laine M, Porola P, Udby L, Kjeldsen L, Cowland JB, Borregaard N, Hietanen J, Stahle M, Pihakari A, Konttinen YT. Low salivary dehydroepiandrosterone and androgen-regulated cysteine-rich secretory protein 3 levels in Sjogren's syndrome. Arthritis Rheum. 2007 Aug;56(8):2575-84. doi: 10.1002/art.22828. PMID 17665393
- [Derived] Virkki LM, Porola P, Forsblad-d'Elia H, Valtysdottir S, Solovieva SA, Konttinen YT. Dehydroepiandrosterone (DHEA) substitution treatment for severe fatigue in DHEA-deficient patients with primary Sjogren's syndrome. Arthritis Care Res (Hoboken). 2010 Jan 15;62(1):118-24. doi: 10.1002/acr.20022. PMID 20191499